CLINICAL TRIAL: NCT03594903
Title: Maintenance (vs. Change) of Critical Attitudes Towards Psychotherapy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Philipps University Marburg (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 2018-19k
Record Dates: First submitted 2018-07-05; First posted 2018-07-20 (Actual); Last update posted 2018-11-08 (Actual); Status verified 2018-11

CONDITIONS: Negative Therapy Expectation
Keywords: therapy expectation; therapy motivation; critical attitudes towards psychotherapy; expectation violation; Violex model; psychological online-experiment

STUDY DESIGN:
Intervention Model Description: participants are assigned to one of two groups in parallel for the duration of the study
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Expectation violation (positive outcome of therapy) (Experimental): Experimental: patients' report about therapy outcome Video with patients giving information about (mostly) positive therapy outcome
  Interventions: Behavioral: video intervention (therapy expectation violation)
- Control group (symptoms + expectation) (Other): Control group: patient´s report about symptoms and therapy expectations
  Participants in the control group are watching a video with the same patients (actors) as in the experimental video. In this video patients are shown before or after the first therapy session. They are giving information about symptoms and their expectation on therapy but NOT about therapy outcome.
  Interventions: Behavioral: video intervention (symptoms+ expectation)

INTERVENTIONS:
Behavioral: video intervention (therapy expectation violation) — The investigators asked experts (psychotherapist and scientists in the area of clinical psychology) about typical therapy expectation violations in therapy and searched the literature for information about typical therapy processes and outcomes. Having these information they designed a script for the experimental video. The patients in the video are played by actors aged from 28 to 58 years (two male and two female actors). Patients are representing common mental disorders (depression, anxiety disorder, alcohol addiction, depression after physical disease). The abbreviated name, age and disorder of the patients is displayed for 3 seconds in the video. The patients are giving information about the mostly positive outcome and the process of their therapy. All participants are watching a video with all patients (7 minutes). The videos (control and experimental group) have been evaluated by 12 experts (psychotherapist and scientists in the area of clinical psychology).
  Arms: Expectation violation (positive outcome of therapy)
Behavioral: video intervention (symptoms+ expectation) — Participants in the control group are watching a video with the same patients (actors) as in the experimental video. In this video patients are shown before or after the first therapy session. They are giving information about symptoms and their expectation on therapy but NOT about therapy outcome.
  Arms: Control group (symptoms + expectation)

SUMMARY:
The aim of the study is to evaluate the effectiveness of a video intervention, which was designed to improve therapy expectation of persons with critical attitudes towards psychotherapy via violating their expectations about therapy. Therefore, 120 participants will be recruited and randomized to two groups:

(1) An experimental group that is watching a video with patients (actors) that are giving oral information about their therapy and the mostly positive therapy outcome, (2) a control group that is watching a video with the same patients before therapy or after the first therapy session who are giving information about symptoms and their expectation on therapy. The primary outcome is the Milwaukee Psychotherapy Expectation Questionnaire (MPEQ) collected before and after the video.

DETAILED DESCRIPTION:
Therapy expectation is one of the main predictors of therapy outcome. This could be shown through many results in the medical sector as well as in studies that are focusing on psychotherapeutic interventions across different mental disorders. Although psychotherapy is a successful treatment for many disorders it is still hold in low esteem by some parts of the population and from some patient groups in particular. This can cause (that) patients who are in need of treatment not being recommended to the right therapy. Furthermore patients with low therapy expectation are more likely to (prematurely) abandon their therapy or having a lower therapy outcome. So therapy expectation should definitely be addressed in the very first therapy sessions because of it´s high impact.

The Violex-model gives an overview on how expectations in general are developed, maintained or modified. The model postulates that a process called immunization can lead to maintenance of expectation even if they receive information that contradicts their expectation. However no trial has yet examined weather the suggestions of the model are adaptable to therapy expectation. Therefore the investigators are recruiting participants with critical attitudes towards psychotherapy and trying to provoke expectation violation via an online experiment containing videos with patients reporting about their mostly positive outcome of psychotherapy. A control group is watching a video with patients who are just giving information about their symptoms and their first impressions on psychotherapy. The primary outcome is the Milwaukee Psychotherapy Expectation Questionnaire (MPEQ) collected before and after the video. Furthermore the participants are asked about their attitudes towards psychotherapeutic treatment (QAPT, German Version FEP), their own experience with psychotherapy and experiences of relevant others, behavioral intensions towards seeking psychotherapy, their mental wellbeing and demographic data. Before watching the video participants are also asked to formulate one to three individual expectations on psychotherapy. After watching the video they are asked how much they still believe in their individual expectation.

The investigators are aiming to modify low therapy expectation by generating expectation violation and paying particular attention to the issue of persistence of expectations via having a closer look on possible immunization strategies. For doing so they developed immunization items (data- and construct-orientated) that are shown at the end of the experiment.

ELIGIBILITY:
Inclusion Criteria:

* Age: 18 years or older
* Critical attitude towards psychotherapy (self-selection)
* ability to speak and read German
* access to the internet

Exclusion Criteria:

* known major mental disorder, such as schizophrenia or another psychotic disorder, or drug or alcohol addiction or dementia (based on self-report)
* medication that influences cognitive processes substantially (benzodiazepine)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2018-11 (Estimated); Primary Completion 2019-01 (Estimated); Study Completion 2019-01 (Estimated)

PRIMARY OUTCOMES:
Milwaukee Expectation Questionnaire (MPEQ) | changes from baseline to after watching the video (approx. 20 minutes later)
  Therapy expectation measured by the Milwaukee Expectation Questionnaire (MPEQ) - 13 items, German translation, self-report, subscales: process expectation and outcome expectation, total mean from min. 0 to max.10.

SECONDARY OUTCOMES:
FEP/ QAPT | changes from baseline to after watching the video (approx. 20 minutes later)
  Self-report measure of attitudes towards psychotherapeutic treatments FEP (Fragebogen zu Einstellungen gegenüber der Inanspruchnahme psychotherapeutischer Hilfe) / Attitudes towards Psychotherapeutic Treatment (QAPT); total score from min. 11 to max. 44
Self-report of individual expectations towards psychotherapy; mean from min. 1 to max. 7 | changes from baseline to after watching the video (approx. 20 minutes later)
Self-report of behavioral intensions towards seeking psychotherapy (self-developed items); mean from min. 1 to max.7 | changes from baseline to after watching the video (approx. 20 minutes later)

OTHER OUTCOMES:
Brief symptom inventory (BSI-18); total score from min.0 to max. 72 | Baseline
  moderator
Self-report measure of own experiences with psychotherapy, reports of experiences with psychotherapy of relevant others and perceived cultural reputation of psychotherapy; single scores from min 1. to max. 5. | Baseline
  moderator
Self-report of possible immunization strategies while or after watching the video (data- and concept-orientated); mean from min. 1 to max. 5 | After watching the video (approx. 20 minutes after baseline)
  moderator
Self-report of perceived sympathy, attractiveness, friendliness and identification with the patients in the video; single scores from min. 1 to max. 5 | After watching the video (approx. 20 minutes after baseline)
  moderator

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Braun-Koch K, Rief W. Maintenance vs. Change of Negative Therapy Expectation: An Experimental Investigation Using Video Samples. Front Psychiatry. 2022 Apr 4;13:836227. doi: 10.3389/fpsyt.2022.836227. eCollection 2022. PMID 35444567